CLINICAL TRIAL: NCT00258973
Title: Office Practice Assessment of Carotid Atherosclerosis Using Handheld Ultrasound (OPACA) Study
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: M-2005-1281
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Atherosclerosis
Keywords: Hand held Ultrasound; Office practice; Atherosclerosis prevention; Ultrasound training
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Carotid Ultrasound performed in office practice

SUMMARY:
The purposes of this study are to determine:

1. Inter-site variability in CIMT image measurement using SonoCalcTM.
2. If non-sonographer health care professionals working in an office practice setting can be trained to follow a carotid scanning protocol that permits (a) accurate measurement of CIMT and (b) determination of plaque presence.
3. If (a) CIMT measurements and (b) determination of plaque presence by non-sonographer health care professionals are bioequivalent to those made by a core laboratory.
4. If CIMT measurements and plaque assessment performed in office practices lead to meaningful changes in patient and physician behavior related to cardiovascular disease prevention.

DETAILED DESCRIPTION:
Phase

IV

Type (observational vs. interventional)

Observational

Currently recruiting or not?

NO

Randomized? (or not)

No Blinded? (single, double, or open)

Primary outcome(s)

Bioequivalency of carotid IMT measurements.

Secondary outcome(s)

Variability in carotid IMT measurements Intention to behavior change in patients Effects of carotid IMT on physician management

Type of Intervention (e.g., drug; device; behavioral)

Device

Name of Intervention

Handheld ultrasound measurement of carotid IMT

ELIGIBILITY:
Inclusion Criteria:

* Males over 45 years and females over 55 years of age with at least one additional risk factor for coronary artery disease.
* Females 45-54 years old may be enrolled if they have a family history of CHD (myocardial infarction, coronary artery bypass graft surgery, angioplasty, sudden cardiac death) in a male first degree relative <55 or a female first degree relative <65 years old AND at least one additional risk factor for coronary artery disease.

Exclusion Criteria:

* Age >70 years
* Subjects taking cholesterol-lowering medications
* Active liver disease
* Active thyroid disease
* Uncontrolled hypertension
* Chronic kidney disease
* History of coronary artery disease
* History of cerebrovascular disease
* History of peripheral arterial disease

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2006-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalency of carotid IMT measurements.

SECONDARY OUTCOMES:
Variability in carotid IMT measurements
Intention to behavior change in patients
Effects of carotid IMT on physician management

CONTACTS AND LOCATIONS:
Overall Officials: James Stein, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States